CLINICAL TRIAL: NCT02879214
Title: Simultaneously Integrated Dose Escalation for Locally Advanced Cervical Cancer (SIDE, Advanced Squamous Cervical Cancer Trial)
Brief Title: Simultaneously Integrated Dose Escalation for Locally Advanced Cervical Cancer
Acronym: Side
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, ming zeng, MD, Director of Cancer Center, Sichuan Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201604
Record Dates: First submitted 2016-08-10; First posted 2016-08-25 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Squamous Cell Carcinoma of Cervix
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SIDE cervical trial (Experimental): To Maximal downstage locally advanced squamous cell cervical cancer before minimal invasive surgical resection. The SIDE study is to use both RT dose escalation to the biological target defined by PET and Chemo dose escalation composited with two drugs to achieve maximal reduction of tumor burden, providing feasibility of minimal invasive surgical resection.
  Interventions: Radiation: Simultaneous boost along with chemo

INTERVENTIONS:
Radiation: Simultaneous boost along with chemo — Prior studies have utilized a sequential boost to deliver a total dose of 55 - 60 Gy to the pelvic sidewall (covering the lower pelvic lymph nodes), including 8-10 Gy that is usually delivered with brachytherapy (1-3), the studies often use single drug. This study treatment plan will use dose intensify in both chemotherapy and radiation. The chemotherapy have two drugs regimens of mitomycin with cisplatin or taxol with cisplatin along of radiation dose escalate, the RT dose escalation to biological GTV defined by PET scan to dose of 57.50 Gy in 25 fx while the elective volumes are held constant at 45 Gy.

SUMMARY:
The purpose of this study is to determine the feasibility of minimal invasive surgical resection through simultaneously integrated dose escalation given concurrently with chemotherapy for locally advanced squamous cell cervical cancer.

DETAILED DESCRIPTION:
Concurrent radiation therapy and chemotherapy is the standard of care for locally advanced cervical cancer. While there are several acceptable means to boost the disease in the low pelvis (i.e. brachytherapy, IMRT, or external beam), there is limited research into minimal invasive surgical resection after maximal downstage. This protocol is designed to determine the dose escalation of both chemo and radiation for treating tumor bearing regions within the abdomen and pelvis, using an two drug chemotherapy in first cycle of mitomycin/cisplatin or taxol/cisplatin along with simultaneously integrated boost technique to Biological target area defined by PET scan. This dose escalation is to downstage disease for minimal invasive surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed squamous cell carcinoma of cervix, able to receive chemotherapy and concurrent chemoradiotherapy.

Good performance status. Negative pregnancy test in women of child-bearing potential. Signed study-specific informed consent. Lab results within study specific limits

Exclusion Criteria:

* Prior radiation to the abdomen or pelvis. A history of Scleroderma or Inflammatory bowel disease. Contraindication to chemotherapy or radiation

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
To observe the efficacy from radiation therapy dose escalation | 4 year
  40 participants will be evaluated with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
To evaluate the chemoradiation in Stage IIB~ III carcinoma cervix | 4 years
  40 Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0, to see any adverse events within 12 months
Disease free survival(DFS) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zeng, MD PhD, Study Chair — Sichuan Provincial People Hospital, Sichuan Academy of Medical Sciences
Locations (1):
- Sichuan PPH, Departmentn of Gynecology Oncology, Chengdu, Sichuan, China